CLINICAL TRIAL: NCT01945008
Title: Prospective Multicentric Observational Study in HCV Chronic Infected Patients.
Brief Title: Observational Study in HCV Chronic Infection
Status: Completed | Type: Observational
Sponsor: Istituto Superiore di Sanità (Other)
Responsible Party: Principal Investigator, Stefano Vella, Director of the Department of Therapeutic Research and Medicines Evaluation, Istituto Superiore di Sanità
Other Study IDs: PITER 01
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Hepatitis C, Chronic
Keywords: HCV; observational study; HCV direct-acting antiviral agents
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatitis-C infected patients: Patients with Hepatitis-C infection untreated at the enrolment

SUMMARY:
HCV infection is the most frequent cause of liver chronic disease, cirrhosis and hepatocellular carcinoma in western countries.

To date, the standard antiviral treatment, including pegylated interferon (PEG-IFN) plus ribavirin (RBV), has relatively low effectiveness in patients infected with genotype 1 and 4, and is associated with important adverse side effects, that lead to treatment interruption in approximately 30% of cases.

The recent association of first generation HCV- specific direct-acting antiviral agents (DAAs) (telaprevir and boceprevir) to standard treatment has resulted in higher SVR rates, also in patients infected with genotype-1 HCV and in non responders to PEG-IFN plus RBV. While several new DAAs are in development, the ultimate goal is represented by IFN-free regimens, that will provide a great advantage in terms of patients adherence to therapy and quality of life.

In this context, prospective observational studies are needed to evaluate the real and long-term impact of the new DAAs in the clinical practice, in terms of efficacy, safety, costs and impact on patients quality of life.

Italy is the European country with the greatest number of HCV infected people (average, 3% of population), with higher prevalence in the center and in the south of the country, especially in older individuals, and the highest mortality caused by hepatocellular carcinoma. Genotype 1 is the most frequent one (in more than 50% of infected people). DAAs were approved at the end of 2012. For these reasons, Italy represents an interesting context for collecting data on long-term efficacy, safety and tolerability of new anti-HCV treatments.

The PITER cohort study, developed in the frame of Italian Platform for the study of the therapy of viral hepatitis a prospective observational study, is based on a large cohort of HCV infected patients from more than 100 clinical centers distributed on the whole national area.

The main aims of the PITER longitudinal cohort study are: 1) to produce of an ongoing and continuously updated picture of the changing epidemiology of HCV infection in the country; 2) to evaluate in a real-life setting the expected impact of DAAs on the natural course of infection and on long-term morbidity and mortality.

DETAILED DESCRIPTION:
Collected data will include clinical, laboratory and anatomopathological information and will be recorded in electronic CRF, at the enrollment and follow-up visits.

Special attention will be devoted to specific patient categories (with HIV, HBV, HDV and HEV coinfections, comorbidities, disease patients who presents signs of liver disease progression). Subjects starting an antiviral regimen will be followed according to specific guidelines.

A sub-study on quality of life/adherence to treatment/treatment satisfaction will be also conducted on all treated patients of the cohort.

ELIGIBILITY:
Inclusion Criteria:

- All HCV infected patients who will consecutively come to the participating clinical centers in a given time span (enrollment periods)

Exclusion Criteria:

* Younger than 18 years
* Patients treated at the moment of the enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient characteristics: :
  * any clinical and histopathologic stage of HCV infection
  * infected by any HCV genotypes
  * Untreated at the time of the enrolment (previously treated subjects are eligible)
  * With/without HBV co-infection
  * With/without HIV co-infection (in any clinical stage of HIV infection, with or without antiretroviral treatment)
Sampling Method: Probability Sample
Enrollment: 7600 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Age distribution at recruitment | ten years
  Age distribution will be expressed in years and reported as median
Sex distribution at recruitment | ten years
  The sex distribution (males and females) will be reported as frequencies (percent)
BMI distribution at recruitment | ten years
  The BMI (kg/m^2) will be expressed in the following cathegories: Underweight, Normal, Overweight, Obese and will be reported as frequencies (percent)
Genotype distribution at recruitment | ten years
  Genotype distribution will be expressed in the following categories: 1 non subtyped, 1a, 1b, 2, 3, 4-5, and will be reported as frequencies (percent)
Liver disease stage at recruitment | ten years
  The liver disease stage distribution will be expressed in the following chategories: F0-F3, F4-cirrhosis, decompensated cirrhosis, HCC, liver transplant, and will be reported as frequencies (percent)
Sustained virological response (SVR) in treated patients | ten years
  Rates of SVR for each expected combination of DAAs used; identification of factors influencing HCV treatment response in the real life.
Changes in the severity of liver disease | ten years
  Changes in liver function will be evaluated in terms of Child Pugh (C-P) score increase or decrease by 1 or more points, whatever occurred first after the end of treatment.
  This outcome will be expressed as proportions (percent)
Incidence of Hepatocellular carcinoma (HCC) | ten years
  Incidence of HCC will be evaluated on the basis of the first diagnosis reported after the end of treatment, excluding prevalent HCC cases occurred before treatment.
  Cumulative incidence will be expressed as proportions (percent)
Incidence and recurrence of decompensated cirrhosis | ten years
  Liver decompensating event is defined as the presence or appearance of ascites and/or portal hypertensive gastrointestinal bleeding and/or hepatic encephalopathy.
  Incidence of a decompensating event will be evaluated on the basis of the first occurrence after the end of treatment, excluding cases occurred before treatment.
  Recurrence of decompensation will be evaluated on the basis of the first events in patients with previous history of decompensated cirrhosis.
  Cumulative incidence or recurrence will be expressed as proportions (percent)

CONTACTS AND LOCATIONS:
Overall Officials: Loreta Kondili, MD, Principal Investigator — Istituto Superiore di Sanità
Locations (1):
- Istituto Superiore di Sanità, Rome, Italy